CLINICAL TRIAL: NCT07159685
Title: Sex-Based Differences of Left Atrium: Impact on Atrial Fibrillation Ablation.
Brief Title: Sex-Based Differences of LA: Impact on AF Ablation.
Status: Not yet recruiting | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Chief of Electrophysiology Unit, Centro Medico Teknon
Other Study IDs: Sex-Tailored By-LAWT AF
Record Dates: First submitted 2025-08-13; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent a first ablation procedure for paroxysmal or persistent atrial fibrillation: patients who underwent a first ablation procedure for paroxysmal or persistent atrial fibrillation
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Atrial fibrillation ablation with RF, guided by navigation system

SUMMARY:
The aim of the study is to assess sex-related differences in patients who underwent a first ablation procedure for paroxysmal or persistent AF, guided by the personalized ablation strategy of the BY-LAWT protocol. Specifically, to compare anatomical characteristics, procedural parameters, and clinical outcomes between sexes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a first ablation procedure for atrial fibrillation (paroxysmal or persistent).
* Availability of an adequate pre-procedural cardiac CT scan for LAWT, LAV and inFAT analysis.
* Availability of complete procedural data, including ablation index (AI) values recorded using the SmartTouch catheter (Biosense Webster).
* Availability of 12-month follow-up data for efficacy and safety endpoint evaluation.
* Ablation performed according to the by-LAWT protocol

Exclusion Criteria:

* Age < 18 years.
* Previous cardiac ablation (including AF ablation or other arrhythmias).
* Incomplete data regarding procedural parameters, or follow-up.
* Poor quality pre-procedural cardiac MDCT
* Ablation not performed according to the BY-LAWT protocol.
* Structural heart disease (e.g., dilated cardiomyopathy, valvular heart disease with surgical indication) that could substantially influence atrial dimensions or ablation response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent a first ablation procedure for paroxysmal or persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy in AF freedom | from the procedure to 12 months later
  The primary efficacy endpoint will be freedom from any atrial arrhythmia (AF, atrial tachycardia [AT], or atrial flutter [AFL]) at the 12-month follow-up. The following definitions apply

CONTACTS AND LOCATIONS:
Locations (1):
- Teknon Medical center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT07159685/Prot_SAP_ICF_000.pdf